CLINICAL TRIAL: NCT02884908
Title: Pharmacogenetic Treatment With Anti-Glutaminergic Agents for Comorbid PTSD & AUD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Melanie E Bennett, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00069465; 5R01AA024760 (NIH)
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Results first posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: PTSD; Alcohol Use Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Pregabalin + BBCET - NI/I/II type (Experimental): This group will be comprised of subjects with the NI/I/II type who receive study medication (Pregabalin) and Brief Behavioral Compliance Enhancement Treatment (BBCET).
  Interventions: Drug: Pregabalin plus BBCET
- Pregabalin + BBCET - NI/NI type (Experimental): This group will be comprised of subjects with the NI/NI type who receive study medication (Pregabalin) and Brief Behavioral Compliance Enhancement Treatment (BBCET).
  Interventions: Drug: Pregabalin plus BBCET
- Placebo + BBCET - NI/I/II type (Placebo Comparator): This group will be comprised of subjects with the NI/I/II type who receive placebo and Brief Behavioral Compliance Enhancement Treatment (BBCET).
  Interventions: Other: Placebo plus BBCET
- Placebo + BBCET - NI/NI type (Placebo Comparator): This group will be comprised of subjects with the NI/NI type who receive placebo and Brief Behavioral Compliance Enhancement Treatment (BBCET).
  Interventions: Other: Placebo plus BBCET

INTERVENTIONS:
Drug: Pregabalin plus BBCET — Medication; BBCET = Brief Behavioral Compliance Enhancement Treatment
  Other Names: Lyrica
  Arms: Pregabalin + BBCET - NI/I/II type; Pregabalin + BBCET - NI/NI type
Other: Placebo plus BBCET — Placebo; BBCET = Brief Behavioral Compliance Enhancement Treatment
  Arms: Placebo + BBCET - NI/I/II type; Placebo + BBCET - NI/NI type

SUMMARY:
The primary study objective is to determine the efficacy of pregabalin administered orally for a period of 12 weeks in reducing risky drinking and symptoms of posttraumatic stress disorder who have selected genotypes at the gamma-amino butyric acid transporter and receptor genes. The secondary objective is to assess the safety and tolerability of pregabalin in participants with alcohol use disorder and co-occurring posttraumatic stress disorder who have selected genotypes at the gamma-amino butyric acid transporter and receptor genes. The investigators will utilize a sample of African-Americans that includes both genders and individuals with different types of trauma.

DETAILED DESCRIPTION:
Nearly 60% of individuals with posttraumatic stress disorder (PTSD) have a comorbid alcohol use disorder (AUD). This comorbidity is associated with more severe PTSD symptoms, higher rates of psychosocial and medical problems, higher relapse rates, and poorer treatment outcome. Pre-clinical studies have indicated that PTSD and AUD share common molecular underpinnings. Particularly, the adaptations in the brain neurotransmitter systems to chronic excessive drinking that are evident during alcohol withdrawal share similarities with PTSD cluster B and E symptoms (characterized by symptoms of re-experiencing and hyper-arousal), which initiate a cycle of relapse into excessive drinking and worsening of PTSD symptoms. Excessive glutamate and reduced gamma-amino butyric acid (GABA) neurotransmitter concentrations were found in various brain regions in individuals with co-morbid PTSD/AUD. The anticonvulsant pregabalin (with high affinity for the alpha-2-delta auxiliary site of voltage gated calcium channels) that modulates the effects of the GABA transporter (GAT-1) and increases its density of GABA, has shown preliminary efficacy in reducing drinking in AUD with comorbid generalized anxiety disorder, and improves outcomes from PTSD. Large scale studies with ample statistical power in VA settings and community populations, with diverse combat and non-combat related trauma, are now warranted to evaluate the promising preliminary evidence that pregabalin can improve outcomes for those with AUD and PTSD. An important personalized medicine approach to optimize pregabalin efficacy would be to select individuals with AUD and PTSD with genetic variation at the GAT-1 transporter so as to match its potential therapeutic effects with specific types of individual. In African-Americans, variants at the SLC6A1 gene promoter region insertion (i.e., non-insertion/insertion or insertion/insertion (NI/I or I/I) compared with those of Non-insertion/Non-insertion (NI/NI) type have significantly higher levels of GAT-1promoter activity. The investigators will, therefore, segregate our target sample by genetic variation at the GAT-1 transporter. Because of the low allelic frequency of individuals with the double copy insertion, the investigators will combine these into one group with those with the single copy (i.e., NI/I/II).

This study will test the efficacy of pregabalin in reducing both alcohol consumption and PTSD symptoms in 2 treatment groups of medication (pregabalin 450 mg/day and placebo) x 2 genetic variants (NI/I/II vs. NI/NI) in a double- blind, placebo-controlled 14-week clinical trial (screening, 12 weeks of study medication, follow-up call). After a one-week screening period, pregabalin dose (and placebo) will be titrated to the target dose from baseline to week 3 using a double-dummy procedure to ensure equivalence of capsules received. The investigators will utilize a sample of African-American participants with co-occurring AUD and PTSD that includes both genders and individuals with different types of trauma. Participants will receive standardized discussions to enhance compliance with study medication at all visits. The specific aims are:

Specific Aim 1: Independent of race, to test the hypothesis that AUD/PTSD participants treated with pregabalin will demonstrate a greater reduction in heavy drinking than placebo treated participants.

Specific Aim 2: Independent of race, to test the hypothesis that AUD/PTSD participants treated with pregabalin will demonstrate a greater reduction in PTSD cluster B or E symptoms (or both) than placebo-treated participants.

Specific Aim 3: To test the hypothesis that race will moderate the effects of pregabalin examined in Aims 1 and 2.

Specific Aim 4: To test the hypothesis that the treatment responses to pregabalin specified in Aims 1 and 2 are modulated by genetic variations within SLC6A1 gene in AUD/PTSD in both African American and European American populations.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of self-reported European or African American ancestry who have given written informed consent
2. Age 18 to 65 years and weighing within 30% of their ideal body weight (Metropolitan Life Tables). Also, subjects must weigh at least 40 kg and no more than 155 kg.
3. Good physical health as determined by a complete physical examination, an EKG within normal limits, and laboratory screening tests within acceptable parameters (see exclusion criteria)
4. Current Diagnostic and Statistical Manual of Mental Disorders Version 5 (DSM-5) diagnosis of posttraumatic stress disorder (PTSD)
5. Current DSM-5 diagnosis of alcohol use disorder (AUD) of moderate or greater severity (i.e., 4 or more AUD criteria endorsed) in the last 3 months
6. Currently drinking ≥21 alcohol units/week for women and ≥28 alcohol units/week for men in the last 30 days and have met these criteria 7 days prior to randomization.
7. Provide evidence of stable residence in the last month prior to enrollment in the study, and have no plans to move in the next 9 months
8. The pregnancy test for females at intake must be negative. Additionally, women of childbearing potential must be using an acceptable form of contraception. These include: oral contraceptives, hormonal (levonorgestrel) or surgical implants, or barrier plus spermicide.
9. Literate in English and able to read, understand, and complete the rating scales and questionnaires accurately, follow instructions, and make use of the behavioral treatments
10. Express a wish to stop drinking
11. Willing to participate in behavioral treatments for PTSD and AUD

Exclusion Criteria:

1. Any current DSM 5 psychiatric disorder other than PTSD, AUD, or Tobacco Use Disorder that warrants treatment or would preclude safe participation in the protocol
2. Elevation of liver enzymes (SGOT), serum glutamic pyruvic transaminase (SGPT), blood urea nitrogen (BUN), or lactate dehydrogenase (LDH) greater than four times the upper limit of the normal range, or elevated bilirubin
3. Severe alcohol withdrawal symptoms that, in the physician's opinion, require inpatient treatment
4. Serious medical comorbidity requiring medical intervention or close supervision, or any condition that can interfere with the receipt of topiramate
5. Severe or life-threatening adverse reactions to medications in the past or during this clinical trial
6. Female subjects who are pregnant, lactating, or not adhering to an acceptable form of contraception at any time during the study
7. Received inpatient or outpatient treatment for alcohol dependence within the last 30 days
8. Compelled to participate in an alcohol treatment program to maintain their liberty
9. Members of the same household
10. Active tuberculosis
11. Concurrent treatment with any medications having a potential effect on alcohol consumption and related behaviors, or mood. These include: opioid antagonists (e.g., naltrexone), glutamate antagonists (e.g., topiramate or acamprosate), serotonin reuptake inhibitors (e.g., fluoxetine), serotonin antagonists (e.g., ritanserin or buspirone), other antidepressants (e.g., tricyclic antidepressants or monoamine oxidase inhibitors), dopamine antagonists (e.g., haloperidol), calcium channel antagonists (e.g., isradipine), or compounds with actions similar to disulfiram (Antabuse®) or nicotine.
12. Before double-blind randomization, urine positive for opiates, cocaine, amphetamines, barbiturates, benzodiazepines, or prescription or non-prescription drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Following the NIH policy, and the Principles and Guidelines for Recipients of NIH Research Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources, the investigators will provide all of our research resources available for research purposes to qualified individuals within the scientific community after publication of our results.
  Sharing of all of the research resources generated by this funded project will be in accordance with the federal rules or regulations imposed upon by the University of Maryland, Baltimore. The investigators will make the results available in accordance with the NIH Data Sharing policy. The investigators will analyze data and submit for peer reviewed publications in scientific journals. The investigators will also present the data in scientific meetings, symposia, or other scientific communications consistent with academic standards.

REFERENCES:
- [Background] Baldwin DS, Anderson IM, Nutt DJ, Allgulander C, Bandelow B, den Boer JA, Christmas DM, Davies S, Fineberg N, Lidbetter N, Malizia A, McCrone P, Nabarro D, O'Neill C, Scott J, van der Wee N, Wittchen HU. Evidence-based pharmacological treatment of anxiety disorders, post-traumatic stress disorder and obsessive-compulsive disorder: a revision of the 2005 guidelines from the British Association for Psychopharmacology. J Psychopharmacol. 2014 May;28(5):403-39. doi: 10.1177/0269881114525674. Epub 2014 Apr 8. PMID 24713617
- [Background] Baniasadi M, Hosseini G, Fayyazi Bordbar MR, Rezaei Ardani A, Mostafavi Toroghi H. Effect of pregabalin augmentation in treatment of patients with combat-related chronic posttraumatic stress disorder: a randomized controlled trial. J Psychiatr Pract. 2014 Nov;20(6):419-27. doi: 10.1097/01.pra.0000456590.12998.41. PMID 25406046
- [Background] Fowler M, Garza TH, Slater TM, Maani CV, McGhee LL. The relationship between gabapentin and pregabalin and posttraumatic stress disorder in burned servicemembers. J Burn Care Res. 2012 Sep-Oct;33(5):612-8. doi: 10.1097/BCR.0b013e31823dc710. PMID 22210072
- [Background] Guglielmo R, Martinotti G, Clerici M, Janiri L. Pregabalin for alcohol dependence: a critical review of the literature. Adv Ther. 2012 Nov;29(11):947-57. doi: 10.1007/s12325-012-0061-5. Epub 2012 Nov 5. PMID 23132700
- [Background] Johannessen Landmark C. Antiepileptic drugs in non-epilepsy disorders: relations between mechanisms of action and clinical efficacy. CNS Drugs. 2008;22(1):27-47. doi: 10.2165/00023210-200822010-00003. PMID 18072813
- [Background] Martinotti G. Pregabalin in clinical psychiatry and addiction: pros and cons. Expert Opin Investig Drugs. 2012 Sep;21(9):1243-5. doi: 10.1517/13543784.2012.703179. Epub 2012 Jun 24. PMID 22725618
- [Background] Martinotti G, Lupi M, Sarchione F, Santacroce R, Salone A, De Berardis D, Serroni N, Cavuto M, Signorelli M, Aguglia E, Valchera A, Iasevoli F, Di Giannantonio M. The potential of pregabalin in neurology, psychiatry and addiction: a qualitative overview. Curr Pharm Des. 2013;19(35):6367-74. doi: 10.2174/13816128113199990425. PMID 23782139
- [Background] Martinotti G, Di Nicola M, Tedeschi D, Andreoli S, Reina D, Pomponi M, Mazza M, Romanelli R, Moroni N, De Filippis R, Di Giannantonio M, Pozzi G, Bria P, Janiri L. Pregabalin versus naltrexone in alcohol dependence: a randomised, double-blind, comparison trial. J Psychopharmacol. 2010 Sep;24(9):1367-74. doi: 10.1177/0269881109102623. Epub 2009 Apr 3. PMID 19346279
- [Background] Mirijello A, Caputo F, Vassallo G, Rolland B, Tarli C, Gasbarrini A, Addolorato G. GABAB Agonists for the Treatment of Alcohol Use Disorder. Curr Pharm Des. 2015;21(23):3367-72. doi: 10.2174/1381612821666150619091858. PMID 26088121
- [Background] Oulis P, Konstantakopoulos G. Efficacy and safety of pregabalin in the treatment of alcohol and benzodiazepine dependence. Expert Opin Investig Drugs. 2012 Jul;21(7):1019-29. doi: 10.1517/13543784.2012.685651. Epub 2012 May 9. PMID 22568872
- [Background] Oulis P, Konstantakopoulos G. Pregabalin in the treatment of alcohol and benzodiazepines dependence. CNS Neurosci Ther. 2010 Spring;16(1):45-50. doi: 10.1111/j.1755-5949.2009.00120.x. PMID 20070788
- [Background] Pae CU, Marks DM, Han C, Masand PS, Patkar AA. Pregabalin augmentation of antidepressants in patients with accident-related posttraumatic stress disorder: an open label pilot study. Int Clin Psychopharmacol. 2009 Jan;24(1):29-33. doi: 10.1097/YIC.0b013e32831feea9. PMID 19060720
- [Background] Shorter D, Hsieh J, Kosten TR. Pharmacologic management of comorbid post-traumatic stress disorder and addictions. Am J Addict. 2015 Dec;24(8):705-12. doi: 10.1111/ajad.12306. Epub 2015 Nov 20. PMID 26587796
- [Background] Strawn JR, Dowling BP, Geracioti TD Jr. Pregabalin treatment of posttraumatic stress disorder. J Clin Psychopharmacol. 2008 Oct;28(5):596-7. doi: 10.1097/JCP.0b013e318184c8f2. No abstract available. PMID 18794673
- [Derived] Wheeler PB, Mackey CD, Moskal D, Brady DJ, Foster KT, Marks RM, Dickerson DL, Kelly DL, Bennett ME, Roche DJO. Religiosity and the relationship between sexual trauma, alcohol use, and sleep quality: a moderated mediation model. Alcohol Alcohol. 2025 May 14;60(4):agaf030. doi: 10.1093/alcalc/agaf030. PMID 40483726
- [Derived] Moskal D, Bennett ME, Marks RM, Roche DJO. Associations among Trauma Exposure, Post-Traumatic Stress Symptoms and Alcohol Use in Black/African American Treatment-Seeking Adults. J Dual Diagn. 2024 Jan-Mar;20(1):5-15. doi: 10.1080/15504263.2023.2286025. Epub 2024 Feb 1. PMID 38113919
- [Derived] Marks RM, Bennett ME, Williams JBW, DuMez EL, Roche DJO. SIGH, what's in a name? An examination of the factor structure and criterion validity of the (Structured Interview Guide for the) Hamilton Anxiety scale (SIGH-A) in a sample of African American adults with co-occurring trauma experience and heavy alcohol use. Exp Clin Psychopharmacol. 2022 Dec;30(6):841-852. doi: 10.1037/pha0000508. Epub 2021 Jul 22. PMID 34291990

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial took place at University of Maryland School of Medicine. Participants were from Baltimore and surrounding counties. The study ran 7/17-6/19 when the research center closed. Recruitment resumed 7/19-3/20 when it stopped due to the pandemic. Recruitment resumed 10/20-12/21 with a 1-month stoppage in 1/21 due to the pandemic.
Pre-assignment Details: N=152 signed consent. Of these, 57 were randomized: 32 to pregabalin, 25 to placebo. 94 were not randomized: 1) did not meet alcohol use disorder criteria; 2) did not meet criteria for PTSD or other trauma disorder; 3) did not meet other eligibility criteria.
Groups:
- Pregabalin + BBCET: This group will be comprised of subjects with the NI/I/II type who receive study medication (Pregabalin) and Brief Behavioral Compliance Enhancement Treatment (BBCET).
  Pregabalin plus BBCET: Medication; BBCET = Brief Behavioral Compliance Enhancement Treatment
- Placebo + BBCET: This group will be comprised of subjects with the NI/I/II type who receive placebo and Brief Behavioral Compliance Enhancement Treatment (BBCET).
  Placebo plus BBCET: Placebo; BBCET = Brief Behavioral Compliance Enhancement Treatment
Period: Overall Study
Arm/Group | Pregabalin + BBCET | Placebo + BBCET
Started (Total randomized.) | 32 | 25
African American | 30 | 24
Took 1 Dose of Study Medication | 26 | 18
Completed (Completed 12-week assessment) | 19 | 7
Not Completed | 13 | 18
Not completed — Lost to Follow-up | 13 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin + BBCET | Placebo + BBCET | Total
Number analyzed (Participants) | 32 | 25 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (11.0) | 42.5 (13.0) | 43.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 18 | 13 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 32 | 24 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 24 | 54
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Diagnostic and Statistical Manual 5 (DSM5) Alcohol Use Disorder (AUD) severity [Mean (Standard Deviation); unit: Number of AUD symptoms] — Number of DSM5 AUD symptoms assessed.
  Number of AUD symptoms | 7.8 (2.3) | 8.3 (1.7) | 8.0 (2.1)
Heavy drinking days in the last 30 days [Mean (Standard Deviation); unit: days] | 10.3 (13.2) | 9.9 (11.4) | 10.2 (12.4)
PTSD Cluster B Symptoms (last week) [Mean (Standard Deviation); unit: Number of symptoms] — PTSD Cluster B Symptoms as measured by the PTSD checklist (PCL)
  Number of symptoms | 9.5 (4.7) | 9.8 (4.2) | 9.7 (4.5)
PTSD Cluster E Symptoms (last week) [Mean (Standard Deviation); unit: Number of symptoms] — PTSD Cluster E Symptoms as measured by the PTSD checklist (PCL)
  Number of symptoms | 11.5 (5.6) | 13.1 (4.3) | 12.2 (5.1)

OUTCOME MEASURES:

1. Primary Outcome: Heavy Drinking Days as Measured by the Time Line Follow Back (TLFB)
Description: Heavy drinking days will be derived from the data collected by the TLFB interview for the last 7 days.
Time Frame: 12 weeks
Population: 44 took at least 1 dose of study medication: 26 in the experimental condition and 18 in the placebo condition. This is the analysis population. For some outcomes, there was missing data at the 12-week assessment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pregabalin + BBCET | Placebo + BBCET
Number analyzed (Participants) | 26 | 18
days
  Baseline | 10.5 (13.1) | 10.2 (11.2)
  12-week assessment: number analyzed (Participants) | 19 | 7
  12-week assessment | 1.1 (2.0) | 1.0 (1.8)
Statistical Analysis 1: Comparison: Pregabalin + BBCET vs Placebo + BBCET; Test type: Superiority — Based on randomization to treatment condition, the model assumed no differences at baseline (any difference was assumed due to random sampling error); p = 0.80, Mixed Models Analysis

2. Primary Outcome: PTSD Cluster B Symptoms as Measured by the PTSD Checklist (PCL)
Description: PTSD Cluster B symptoms assessed during treatment will be derived from the data collected with the PCL.
Time Frame: 12 weeks
Population: 4 took at least 1 dose of study medication: 26 in the experimental condition and 18 in the placebo condition. This is the analysis population. For some outcomes, there was missing data at the 12-week assessment.
Measure: Mean (Standard Deviation); unit: number of symptoms
Arm/Group | Pregabalin + BBCET | Placebo + BBCET
Number analyzed (Participants) | 26 | 18
number of symptoms
  Baseline | 9.7 (4.7) | 9.8 (4.1)
  12-week assessment: number analyzed (Participants) | 19 | 7
  12-week assessment | 3.6 (4.6) | 1.6 (2.2)
Statistical Analysis 1: Comparison: Pregabalin + BBCET vs Placebo + BBCET; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.90, Mixed Models Analysis

3. Primary Outcome: PTSD Cluster E Symptoms as Measured by the PCL
Description: PTSD Cluster E symptoms assessed during treatment will be derived from the data collected with the PCL.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of symptoms
Arm/Group | Pregabalin + BBCET | Placebo + BBCET
Number analyzed (Participants) | 26 | 18
number of symptoms
  Baseline | 12.2 (5.4) | 13.3 (4.8)
  12-week assessment: number analyzed (Participants) | 19 | 7
  12-week assessment | 6.4 (5.0) | 4.4 (3.9)
Statistical Analysis 1: Comparison: Pregabalin + BBCET vs Placebo + BBCET; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.38, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: SAEs & AEs were assessed at each visit. SAEs required review/determination by study physician. AE determinations made by study staff. SAEs were medical or psychiatric hospitalizations of any duration. AEs were any reports of medical or psychiatric issues made by participants when queried about their health status in the last week or since the last study visit that did not require hospitalization. Adverse Events were monitored/assessed without regard to specific Adverse Event Term.
Arm/Group | Pregabalin + BBCET | Placebo + BBCET
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/26 | 1/18
Other Adverse Events (participants affected / at risk) | 26/26 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregabalin + BBCET (N=26) | Placebo + BBCET (N=18)
Hospitalization (General disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin + BBCET (N=26) | Placebo + BBCET (N=18)
Reports of medical or psychiatric issues (Ear and labyrinth disorders) | 4 | 1
Reports of medical or psychiatric issues (Blood and lymphatic system disorders) | 1 | 0
Reports of medical or psychiatric issues (Eye disorders) | 2 | 0
Reports of medical or psychiatric issues (Gastrointestinal disorders) | 7 | 3
Reports of medical or psychiatric issues (General disorders) | 12 | 10
Reports of medical or psychiatric issues (Infections and infestations) | 3 | 2
Reports of medical or psychiatric issues (Metabolism and nutrition disorders) | 3 | 2
Reports of medical or psychiatric issues (Nervous system disorders) | 4 | 2
Reports of medical or psychiatric issues (Psychiatric disorders) | 4 | 1
Reports of medical or psychiatric issues (Renal and urinary disorders) | 1 | 2
Reports of medical or psychiatric issues (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Reports of medical or psychiatric issues (Skin and subcutaneous tissue disorders) | 3 | 1

LIMITATIONS AND CAVEATS:
Sample size calculated for effect size=0.31, attrition=25%, correlation among repeated measures=0.55. With power=0.80 & alpha-level=.05/2=.025, N=198 randomized. Due to interruptions/pandemic, N=57 randomized; final analysis N=44 (26 pregabalin/18 placebo). Re-calculated power based on modified primary analysis, achieved sample size, observed attrition rates (40%), & average correlation among repeated measures. Aim1 effect size=0.67, 2-sided alpha=0.05, power=0.80. Aim2 effect sizes=0.68 & 0.63.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/08/NCT02884908/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT02884908/SAP_001.pdf